CLINICAL TRIAL: NCT06726265
Title: TACTI-004, a Double-Blinded, Randomized Phase 3 Trial in Patients With Advanced/Metastatic Non-Small Cell Lung Cancer (NSCLC) Receiving Eftilagimod Alfa (MHC Class II Agonist) in Combination With Pembrolizumab (PD-1 Antagonist) and Chemotherapy.
Brief Title: Study of Eftilagimod Alfa (Efti) in Combination With Pembrolizumab and Chemotherapy Versus Placebo in Combination With Pembrolizumab and Chemotherapy in Participants With Metastatic Non-Small Cell Lung Cancer (NSCLC) (TACTI-004)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Immutep S.A.S. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TACTI-004; 2024-513621-23-00 (EU CTIS Number); KEYNOTE-F91 (Other: Merck Sharp & Dohme LLC); MK-3475-F91 (Other: Merck Sharp & Dohme LLC); IMP321-P026 (Other: Immutep S.A.S.)
Record Dates: First submitted 2024-12-03; First posted 2024-12-10 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-11

CONDITIONS: Advanced/Metastatic Non-Small Cell Lung Cancer (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — soluble LAG-3 protein, human; Carboplatin; Paclitaxel; Cisplatin; Pemetrexed; pembrolizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- efti + Standard of Care arm (Experimental): Combination of efti, pembrolizumab (KEYTRUDA®) and histology-based platinum doublet chemotherapy
  Interventions: Biological: eftilagimod alfa; Drug: carboplatin plus paclitaxel; Drug: cisplatin or carboplatin + pemetrexed; Biological: pembrolizumab (KEYTRUDA®)
- Placebo + Standard of Care arm (Placebo Comparator): Combination of efti-matching placebo, pembrolizumab (KEYTRUDA®) and histology-based platinum doublet chemotherapy
  Interventions: Drug: carboplatin plus paclitaxel; Drug: cisplatin or carboplatin + pemetrexed; Biological: pembrolizumab (KEYTRUDA®); Other: Placebo

INTERVENTIONS:
Biological: eftilagimod alfa — 30 mg of efti every 2 weeks subcutaneously for the first 6 months, thereafter every 3 weeks for up to 24 months in total
  Other Names: IMP321; LAG-3Ig; efti; eftilagimod alpha
  Arms: efti + Standard of Care arm
Drug: carboplatin plus paclitaxel — For participants with squamous histology for 4 cycles (1 cycle = 3 weeks) as follows: every 3 weeks: carboplatin area under the curve (AUC) 5 or 6 in combination with paclitaxel 175 mg/m2 or 200 mg/m2
Drug: cisplatin or carboplatin + pemetrexed — For participants with nonsquamous histology for 4 cycles (1 cycle = 3 weeks) as follows: every 3 weeks: cisplatin 75 mg/m2 or carboplatin AUC 5 or 6 in combination with pemetrexed 500 mg/m2. After the initial 4 cycles, pemetrexed 500 mg/m2 maintenance therapy will be administered every 3 weeks
Biological: pembrolizumab (KEYTRUDA®) — 200 mg pembrolizumab (KEYTRUDA®) every 3 weeks i.v. for up to approximately 24 months
Other: Placebo — efti-matching placebo every 2 weeks subcutaneously for the first 6 months, thereafter every 3 weeks for up to 24 months in total
  Arms: Placebo + Standard of Care arm

SUMMARY:
The purpose of this study is to compare eftilagimod alfa (efti) in combination with pembrolizumab and chemotherapy versus placebo in combination with pembrolizumab and chemotherapy with respect to overall survival (OS) and progression-free survival (PFS) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) among adults with metastatic non-small cell lung cancer (NSCLC).

Participants will receive either efti plus standard treatment (pembrolizumab and platinum doublet chemotherapy) or placebo plus standard treatment and will be treated for up to 2 years.

DETAILED DESCRIPTION:
TACTI-004 is a double-blinded, randomized phase 3 trial in patients with advanced/metastatic non-small cell lung cancer (NSCLC) receiving eftilagimod alfa (major histocompatibility complex (MHC) class II agonist) in combination with pembrolizumab (programmed cell death protein 1 (PD-1) antagonist) and chemotherapy.

The proposed clinical trial aims to compare the efficacy and to demonstrate the superiority of efti combined with standard of care (SoC, pembrolizumab and histology-based chemotherapy) compared to placebo combined with SoC in programmed death-ligand 1 (PD-L1) unselected population as assessed by:

* Overall survival [OS]
* Progression-free survival [PFS] per RECIST 1.1

The trial is planned to be conducted in countries in Asia, Australia, Europe and North and South America in approximately 175 experienced clinical sites.

ELIGIBILITY:
Inclusion Criteria

Participants may be enrolled if they meet all of the following criteria at screening:

1. Willing to give written informed consent and to comply with the protocol.
2. Histologically- or cytologically-confirmed diagnosis of advanced or metastatic (stage IIIB/C or stage IV) non-small cell lung cancer (NSCLC) not amenable to curative treatment or locally available oncogenic driver mutation-based first-line therapy, treatment naïve for systemic therapy given for advanced/metastatic disease.
3. Archival tumor tissue sample or newly obtained core, or excisional biopsy of a tumor lesion not previously irradiated has been provided. Details pertaining to tumor tissue submission can be found in the Laboratory Manual.
4. Availability of programmed death-ligand 1 (PD-L1) biomarker result from central laboratory, using the Food and Drug Administration (FDA) approved Dako standardized diagnostic test (PD-L1 IHC 22C3 pharmDx).
5. Be ≥ 18 years of age on the day of signing the informed consent.
6. Participants assigned male at birth must follow specific contraception guidelines during and after the trial intervention period. The required contraception duration varies by drug. Participants must refrain from donating sperm and either remain abstinent or use condoms with an additional contraceptive method during intercourse with a nonpregnant partner. Contraceptive measures must adhere to local regulations, with stricter local label requirements taking precedence over the trial's guidelines.
7. A participant of childbearing potential (POCBP) is eligible if they are not pregnant, confirmed by a negative pregnancy test before the first trial dose. They must not breastfeed during the trial or for a defined duration after the last dose of each drug. POCBPs must use highly effective contraception, with low user dependency or long-term abstinence during and after the trial intervention, and refrain from egg donation or storage. The required contraception duration varies by drug. Local contraception regulations must be followed.
8. An Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1 assessed within 7 days before randomization.
9. Expected survival > 3 months.
10. Evidence of measurable disease as defined by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as determined by site.
11. Participants must have recovered from all AEs due to previous anticancer therapies to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0 ≤ Grade 1 or baseline. Participants with CTCAE ≤ Grade 2 neuropathy, alopecia, and elevated transaminases in case of liver metastases may be eligible.
12. Participants who received major surgery prior to trial start must have recovered adequately from the toxicity and/or complications from the intervention prior to starting trial treatment.
13. Participants who are hepatitis B surface antigen (HBsAg) positive are eligible if they have received hepatitis B virus (HBV) antiviral therapy for at least 4 weeks, and have undetectable HBV viral load prior to randomization.
14. Participants with history of hepatitis C virus (HCV) infection are eligible if HCV viral load is undetectable at screening and have completed curative antiviral therapy at least 4 weeks prior to randomization.
15. Human immunodeficiency virus (HIV) infected participants must be on anti-retroviral therapy (ART) and have a well-controlled HIV infection/disease.
16. Adequate organ function.

Exclusion Criteria

Participants are to be excluded from the trial at the time of screening for any of the following reasons:

1. Is expected to require any other form of systemic or localized antineoplastic therapy (other than the trial treatment) while on trial (including maintenance therapy with another agent for NSCLC, radiation therapy, and/or surgical resection).
2. Received prior radiotherapy within 2 weeks of start of trial intervention, or has radiation-related toxicities, requiring corticosteroids.
3. Participants whose tumor harbors any of the following actionable molecular alterations:

   1. Epidermal growth factor receptor (EGFR)-sensitizing (activating) mutation
   2. Anaplastic lymphoma kinase (ALK) gene fusion positive (ALK translocation)
   3. c-ROS oncogene 1 (ROS1) translocation
4. For any indication has received any of the following therapies

   1. within 3 weeks prior to cycle 1 day 1: systemic cytotoxic chemotherapy, targeted small molecule therapy (e.g. kinase inhibitors), biological therapy, any other systemic cancer therapy or had major surgery;
   2. within 4 weeks prior to cycle 1 day 1 has been treated with an investigational agent or has used an investigational device, or is still a participant in the active phase of an investigational trial;
   3. within 6 months prior to cycle1 day 1 received lung radiation therapy of >30 Gray (Gy).
5. Has received any treatment as part of adjuvant, neoadjuvant therapy or definitive chemoradiation for the treatment of NSCLC within 12 months prior to the diagnosis of advanced/metastatic disease.
6. Received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or coinhibitory T-cell receptor (e.g., cytotoxic T-lymphocyte-associated protein 4 (CTLA-4), OX40, CD137) or Lymphocyte Activation Gene 3 (LAG-3) targeting therapy (e.g., anti-LAG-3 antibodies). Prior treatment with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent for nonmetastatic resectable NSCLC (e.g. in the neoadjuvant or adjuvant setting) or following definitive chemoradiation, is allowed as long as therapy was completed at least 12 months before diagnosis of metastatic NSCLC.
7. Prior high-dose chemotherapy requiring hematopoietic stem cell rescue.
8. Known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable (i.e., without evidence of progression) for at least 4 weeks as confirmed by repeat imaging performed during trial screening, are clinically stable and have not required steroid treatment for at least 14 days before the first dose of trial intervention.
9. Active infection requiring parenteral systemic therapy within 4 weeks prior to cycle 1 day 1 and/or significant acute or chronic infection in screening and/or on cycle 1 day 1.
10. Evidence of severe or uncontrolled cardiac disease within 6 months prior to first dose of trial treatment including: myocardial infarction, severe/unstable angina, ongoing cardiac dysrhythmias of NCI CTCAE version 5.0 Grade ≥ 2, atrial fibrillation > Grade 2 not controlled by a pacemaker, coronary/peripheral artery bypass graft, symptomatic congestive heart failure (New York Heart Association (NYHA) III-IV), cerebrovascular accident including transient ischemic attack, or symptomatic pulmonary embolism.
11. History of (noninfectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
12. Has active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed.
13. Diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial intervention.
14. Concurrent active Hepatitis B (defined as HBsAg positive and/or detectable HBV DNA) and Hepatitis C virus (defined as anti-HCV Ab positive and detectable HCV RNA) infection.
15. HIV-infected participants with a history of Kaposi sarcoma and/or Multicentric Castleman Disease.
16. History of allogenic tissue/solid organ transplant.
17. Known additional malignancy that is progressing or has required active treatment within the past 3 years.
18. Has hypersensitivity to eftilagimod alfa and/or pembrolizumab (≥Grade 3) and/or any of its excipients.
19. Has hypersensitivity to any component of planned platinum-based doublet chemotherapy and/or any of its excipients.
20. Received a live or live-attenuated vaccine within 30 days before the first dose of trial intervention. Administration of killed vaccines is allowed
21. Has a life-threatening illness unrelated to cancer.
22. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the participant's participation for the full duration of the trial, or is not in the best interest of the participant to participate, in the opinion of the treating Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 756 (Estimated)
Dates: Start 2025-03-21 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Determination of Overall survival (OS) | Up to approximately 54 months
Determination of Progression free survival (PFS) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) | Up to approximately 54 months

SECONDARY OUTCOMES:
Determination of Objective response rate (ORR) per RECIST 1.1 | Up to approximately 54 months
Frequency of adverse events (AEs) | Up to approximately 27 months
Severity of adverse events (AEs) according to the United States National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), v5.0 | Up to approximately 27 months
Determination of Time to Response (TTR) by RECIST 1.1. | Up to approximately 54 months
Determination of Duration of Response (DOR) by RECIST 1.1. | Up to approximately 54 months
Determination of PFS on next line therapy (PFS2) | Up to approximately 54 months

CONTACTS AND LOCATIONS:
Locations (137):
- New Mexico Oncology Hematology Consultants, Ltd., Albuquerque, New Mexico, United States
- Argentina (3):
  - Centro de Endocrinologia y Diabetes Dr. Raul A. Gutman SRL, Buenos Aires
  - Fundacion Respirar, Buenos Aires
  - Sanatorio Parque - Rosario, Rosario
- Australia (8):
  - Lyell McEwin Hospital, Elizabeth Vale
  - Greenslopes Private Hospital, Greenslopes
  - The Alfred Hospital, Melbourne
  - Tasman Oncology Research Ltd, Southport
  - St John of God Subiaco Hospital, Subiaco
  - Royal Darwin Hospital, Tiwi
  - Calvary Mater Newcastle, Waratah
  - Cancer Care Wollongong Pty Limited, Wollongong
- Austria (2):
  - Landeskrankenhaus-Universitätsklinikum Graz, KLinische Abteilung für Pulmonologie, Graz
  - Vienna General Hospital, Vienna
- Belgium (3):
  - Antwerp University Hospital, Antwerp
  - Algemeen Ziekenhuis Maria Middelares, Ghent
  - Clinique et Maternité Sainte-Elisabeth, Namur
- Brazil (5):
  - Centro Integrado de Oncologia de Curitiba - CIONC, Curitiba
  - Cetus Oncologia Hospital Dia - Belo Horizonte, Horizonte
  - Oncosite - Centro de Pesquisa Clinica Em Oncologia Ltda, Ijuí
  - Hospital Nossa Senhora da Conceicao (HNSC), Porto Alegre
  - Hospital Santa Rita - Vitoria, Vitória
- Bulgaria (5):
  - Multiprofile Hospital for Active Treatment - Dobrich AD, Dobrich
  - Multiprofile Hospital For Active Treatment "Dr. Tota Venkova" AD, Gabrovo
  - MHAT Uni Hospital OOD, Panagyurishte
  - Complex Oncology Center Ruse, Rousse
  - Multiprofile Hospital for Active Treatment Serdika EOOD, Sofia
- Canada (3):
  - Brampton Civic Hospital, Brampton
  - McGill University - Jewish General Hospital (JGH) - Lady Davis Institute for Medical Research, Montreal
  - Unite de recherche clinique du CISSS des Laurentides, Saint-Jérôme
- Chile (2):
  - Centro de Oncologia de Precision, Las Condes
  - Facultad Odontología Unipac, Santiago
- Croatia (4):
  - Klinički Bolnički Centar Osijek, Osijek
  - Klinicka Bolnica Centar - Sestre Milosrdnice - Klinika Za Tumore (University Hospital for Tumors), Zagreb
  - Klinički Bolnički Centar Sestre Milosrdnice, Zagreb
  - Klinički Bolnički Centar Zagreb - Klinika Za Plućne Bolesti Jordanovac, Zagreb
- Georgia (4):
  - High-tech Hospital Med Center, Batumi
  - High Technology Medical Center, University Clinic, Tbilisi
  - Institute of Clinical Oncology, Tbilisi
  - Mardaleishvili Medical Centre, Tbilisi
- Germany (12):
  - Klinikum St. Marien, Amberg
  - HELIOS Klinikum Bad Saarow, Bad Saarow
  - Evangelische Lungenklinik Berlin, Berlin
  - Universitätsklinikum Köln, Cologne
  - Agaplesion Medizinisches Versorgungszentrum - Frankfurt gGmbH, Frankfurt
  - Universitätsklinikum Frankfurt, Frankfurt
  - Krankenhaus Nordwest, Frankfurt am Main
  - Asklepios Fachkliniken München-Gauting, Gauting
  - Krankenhaus Martha-Maria Halle-Dölau, Halle
  - Facharztzentrum Eppendorf, Hamburg
  - Gemeinschaftspraxis für Hämatologie und Onkologie, Münster
  - Robert-Bosch-Krankenhaus, Stuttgart
- Greece (8):
  - General Hospital of Athens "Laiko", Athens
  - Sotiria Chest Diseases Hospital, Athens
  - University of Thessaly- General University Hospital of Larissa, Larissa
  - University of Patras - Rio Regional University Hospital, Pátrai
  - Metropolitan Hospital, Department of Oncology, Piraeus
  - Bioclinic of Thessaloniki, Thessaloniki
  - Interbalkan Medical Center of Thessaloniki, Thessaloniki
  - St. Luke's Hospital S.A., Thessaloniki
- Hungary (2):
  - Debreceni Egyetem Klinikai Központ, Debrecen
  - Tolna Vármegyei Balassa János Kórház, Szekszárd
- India (9):
  - HCG Cancer Centre - Double Road (Bangalore Institute of Oncology (BIO)), Bangalore
  - All India Institute of Medical Sciences (AIIMS) - Bhubaneswar, Bhubaneswar
  - Geri Care Hospital T.Nagar, Chennai
  - Voluntary Health Services Hospital, Chennai
  - Chittaranjan National Cancer Institute, Kolkata
  - Maulana Azad Medical College, New Delhi
  - Sunact Cancer Institute Pvt. Ltd., Thane
  - Regional Cancer Centre Thiruvananthapuram, Thiruvananthapuram
  - Tata Memorial Centre - Mahamana Pandit Madan Mohan Malaviya Cancer Centre, Varanasi
- Ireland (4):
  - Cork University Hospital, Cork
  - Beaumont Hospital, Dublin
  - Mater Misericordiae University Hospital, Dublin
  - Tallaght University Hospital, Dublin
- Italy (8):
  - Azienda Ospedaliera San Giuseppe Moscati, Avellino
  - Centro di Riferimento Oncologico (CRO), Aviano
  - Istituto per la Ricerca e la Cura del Cancro (IRCC) - Istituto di Candiolo, Candiolo
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Istituto Nazionale Tumori (INT) "Fondazione G. Pascale" di Napoli, Napoli
  - Azienda Ospedaliera di Perugia - Ospedale Santa Maria della Misericordia, Perugia
  - Arcispedale Santa Maria Nuova, Reggio Emilia
  - Azienda Ospedaliera Santa Maria di Terni, Terni
- Latvia (2):
  - Latvian Oncology Center, Riga
  - Paula Stradiņa Klīniskā Universitātes Slimnīca, Riga
- Lithuania (2):
  - Hospital of Lithuanian University of Health Sciences Kauno Klinikos, Kaunas
  - Nacionalinis Vezio Institutas, Vilnius
- Malaysia (4):
  - Hospital Tengku Ampuan Afzan, Kuantan
  - Hospital Umum Sarawak - Clinical Research Centre, Kuching
  - Gleneagles Medical Centre - Penang, Pulau Pinang
  - Hospital Pulau Pinang, Pulau Pinang
- Poland (5):
  - Szpital Morski im. PCK (Maritime Hospital) (Gdynskie Centrum Onkologii), Gdynia
  - Przychodnia Lekarska "KOMED", Konin
  - Instytut Medyczny Santa Familia Sp. z o. o. w Łodzi, Lodz
  - IP Clinic Sp. z o.o., Lodz
  - Narodowy Instytut Onkologii im. Marii Skłodowskiej-Curie, Warsaw
- Portugal (6):
  - Hospital Garcia de Orta, EPE, Almada
  - Hospital CUF Descobertas, Lisbon
  - Hospital Lusíadas Lisboa, Lisbon
  - Unidade Local de Saude de Santa Maria, EPE - Hospital Pulido Valente, Lisbon
  - Unidade Local de Saude de Loures - Odivelas, E. P. E., Loures
  - Instituto Português Oncologia do Porto Francisco Gentil, EPE, Porto
- Romania (6):
  - Centrul Medical Medicover Victoria, Bucharest
  - Spitalul Memorial Healthcare International, Bucharest
  - Onco Clinic Consult SA, Craiova
  - OncoLab, Craiova
  - Victoria Hospital - Centrul de Oncologie Euroclinic SRL, Iași
  - Ovidius Clinical Hospital S.R.L., Ovidiu
- Spain (14):
  - Hospital Universitari Germans Trias i Pujol, Badalona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Instituto Oncologico Dr. Rosell - Hospital Universitari Quiron Dexeus Location, Barcelona
  - Hospital Universitario Reina Sofía, Córdoba
  - HM Universitario Sanchinarro, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Regional Universitario de Málaga - Hospital General, Málaga
  - Hospital Universitario Central de Asturias, Oviedo
  - Parc Tauli Hospital Universitari, Sabadell
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital Clínico Universitario "Lozano Blesa", Zaragoza
- Prince of Songkhla University, Hat Yai, Thailand
- Turkey (Türkiye) (11):
  - Adana Medical Park Seyhan Hospital, Adana
  - Adana Sehir Training and Research Hospital, Adana
  - Ankara Universitesi Tip Fakultesi Hastaneleri - Cebeci Hastanesi, Ankara
  - Gulhane Egitim ve Arastirma Hastanesi, Ankara
  - Hacettepe Universitesi Kanser Enstitusu (Hacettepe University Cancer Institute), Ankara
  - Uludağ Üniversitesi Tıp Fakültesi, Bursa
  - Istanbul Oncology Hospital, Cevizli
  - Trakya Universitesi Saglik Arastirma ve Uygulama Merkezi Hastane, Edirne
  - Bahcelievler Memorial Hospital, Istanbul
  - T.C. S.B. Prof. Dr. Suleyman Yalcin Sehir Hastanesi, Istanbul
  - Sakarya Universitesi Tıp Fakultesi Dekanligi, Sakarya
- United Kingdom (3):
  - University Hospitals Birmingham NHS Foundation Trust - New Queen Elizabeth Hospital Birmingham, Birmingham
  - The Royal Surrey County Hospital NHS Foundation Trust, Guildford
  - The Christie NHS Foundation Trust - Christie Hospital, Manchester

REFERENCES:
- [Derived] O'Byrne K, Esteban E, Lee CL, Hegmane A, Volovat C, Lo Russo G, Ziogas D, Atmaca A, Sebastian M, Majem M. A phase III placebo-controlled study of eftilagimod alfa plus pembrolizumab and chemotherapy in metastatic non-small cell lung cancer. Future Oncol. 2025 Dec;21(30):3885-3890. doi: 10.1080/14796694.2025.2597404. Epub 2025 Dec 12. PMID 41383151